CLINICAL TRIAL: NCT01414504
Title: Pneumococcal Conjugate Vaccine Followup: Investigation of Serotype-specific Antibody Persistence and B Cell Memory at Age 3-5 Years Following 23valent Pneumococcal Polysaccharide Vaccine at Age 9 Months in PNG Children Previously Primed With 7valent Pneumococcal Conjugate Vaccine
Brief Title: Pneumococcal Conjugate Vaccine Followup
Acronym: PCVFU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: William Pomat (Other Government)
Collaborators: The University of Western Australia (Other)
Responsible Party: Sponsor-Investigator, William Pomat, Senior Research Fellow, Papua New Guinea Institute of Medical Research
Organization: Papua New Guinea Institute of Medical Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCVFU927
Record Dates: First submitted 2011-08-02; First posted 2011-08-11 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Immune Tolerance
Keywords: pneumococcal,; pneumococcal polysaccharide vaccine,; challenge dose,; hyporesponsiveness,; Papua New Guinea
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine; Predictive Value of Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Neonatal PCV + PPV 9 months (Active Comparator): Group 1: Children receiving 7VPCV at 0-1-2 months of age and PPV at 9 months of age
  Interventions: Biological: Prevenar + PPV
- Infant PCV + PPV at 9 months (Active Comparator): Group 2: Children receiving 7VPCV at 1-2-3 months of age and PPV at 9 months of age
  Interventions: Biological: Infant PCV (Prevenar) + PPV at 9 months
- No PCV + PPV at 9 months (Active Comparator): Group 3: Children who only received PPV at 9 months of age
  Interventions: Biological: No Prevenar + PPV at 9 months
- Control (Active Comparator): Group 4: Children who have not received any previous pneumococcal vaccine
  Interventions: Biological: Control

INTERVENTIONS:
Biological: Prevenar + PPV — 0.5mL dose of Prevenar at 0-1-2 months, 0.5mL Pneumovax at 9 months and 0.1mL Pneumovax at 3-5 yrs
  Arms: Neonatal PCV + PPV 9 months
Biological: Infant PCV (Prevenar) + PPV at 9 months — 0.5mL Prevenar at 1-2-3 months,0.5mL Pneumovax (PPV) at 9 months, 0.1mL Pneumovax at 3-5 yrs
  Other Names: Prevenar; Pneumovax23
  Arms: Infant PCV + PPV at 9 months
Biological: No Prevenar + PPV at 9 months — no Prevenar, 0.5mL Pneumovax at 9 months, 0.1mL Pneumovax at 3-5 yrs
  Arms: No PCV + PPV at 9 months
Biological: Control — control, 0.1mL Pneumovax at 3-5yrs
  Arms: Control

SUMMARY:
Recently, controversy has emerged regarding the role of the 23vPPV in infants due to potential immunological hypo-responsiveness (i.e. a poorer immune response to repeat vaccination). Although previous experience of 23vPPV in children in PNG has demonstrated protective efficacy against acute lower respiratory tract infection, the investigators feel it is a matter of urgency to determine if 23vPPV administration provides elevated antibody concentrations at 3 to 5 years of age, and to ensure the immunological safety of the 23vPPV in infants.

Following consent and eligibility assessment, a baseline blood sample and nose swab will be taken, a 0.1ml dose of 23vPPV will be administered and a follow up blood sample and nose swab will be collected 28 days later. The investigators will also collect data on incidence of ALRI in all study participants by medical record review.

ELIGIBILITY:
Inclusion Criteria:

* PNG Infants aged 3 to 5 yrs of age who participated in previous PNG Neonatal PCV study and received PPV between 9 and 12 months of age, or age- and sex-matched controls who live in the same villages or urban area
* Informed parental/guardian consent

Exclusion Criteria:

* Known HIV infection or other immunosuppressive condition or treatment.
* Prior receipt of 2 doses of pneumococcal polysaccharide vaccine

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Measure serotype-specific antibody persistence in children aged 3-5 years after vaccination with 23vPPV at 9 months of age and compared to unvaccinated controls. | 2yrs
  Children who were previously vaccinated with Pneumovax (23vPPV) at 9 months will be followed up at age 3-5 years of age. They will be given a challenge dose of Pneumovax (0.1mL) and followed up 1 months later. Age matched controls identified from each villages will also be recruited and given a challenge dose of Pneumovax. Serotype-specific antibodies will be measure pre- and post-challenge dose to determine anitbody levels.

SECONDARY OUTCOMES:
Measure the number of circulating serotype-specific memory B-cells pre- & post- booster immunisation | 2yrs
Measure nasopharyngeal pneumococcal serotype-specific carriage rates pre- and post- 23vPPV challenge dose | 2yrs

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Richmond, MD, Principal Investigator — School of Paediatrics and Child Health, University of Western Australia; Deborah Lehmann, MSc, Principal Investigator — Telethon Institute for Child Health Research; William S Pomat, PhD, Principal Investigator — Papua New Guinea Institute of Medical Research
Locations (1):
- PNG Institute of Medical Research, Goroka, Eastern Highlands Province, Papua New Guinea

REFERENCES:
- [Derived] van den Biggelaar AHJ, Richmond PC, Fuery A, Anderson D, Opa C, Saleu G, Lai M, Francis JP, Alpers MP, Pomat WS, Lehmann D. Pneumococcal responses are similar in Papua New Guinean children aged 3-5 years vaccinated in infancy with pneumococcal polysaccharide vaccine with or without prior pneumococcal conjugate vaccine, or without pneumococcal vaccination. PLoS One. 2017 Oct 13;12(10):e0185877. doi: 10.1371/journal.pone.0185877. eCollection 2017. PMID 29028802